CLINICAL TRIAL: NCT01552317
Title: OxCKD1 - a Randomised Controlled Trial of the OxSalt1 Care Bundle to Help Renal Patients Learn How to Lower the Salt Content of Their Diets.
Brief Title: OxCKD1 -Empowering Healthy Lifestyle Choices in Chronic Kidney Disease
Acronym: OxCKD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: British Renal Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OxCKD1
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2014-12

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A package of advice and interventions to help participants reduce their salt intake.
  Interventions: Other: OxSalt care bundle
- Normal care (No Intervention): This group will receive the normal care that they would get anyway.

INTERVENTIONS:
Other: OxSalt care bundle — A care bundle consisting of a range of features to help patients to reduce their salt intake such as reminder emails, phone calls and a website.
  Arms: Intervention

SUMMARY:
Patients with kidney disease benefit from reducing the amount of salt in the food that they eat. The benefits include lower blood pressure and better kidney function. Therefore, lowering the amount of salt that is eaten could reduce the number of people who will develop kidney failure. The effect on blood pressure could also reduce the number of strokes and heart attacks. Similar benefits are also seen for people without kidney disease.

Guidelines for patients with kidney disease recommend that they lower the amount of salt that they eat, but most patients do not manage to do this. The reasons for this are not unclear, but are likely to reflect the difficulty that patients have in reducing the amount of salt in their food and the nature of the advice that they are given.

The investigators have developed a package of interventions to help patients to make healthier choices that will lower their salt intake. The package helps patients to learn about salt in food and how to avoid it. It provide practical advice on cutting down on salt using information booklets, text messages, emails, telephone calls, and a website.

Participants will be recruited from hospital kidney clinics and general practice. The investigators will randomly allocate participants to receive either the normal care that they would get or to receive the new package of interventions to help them lower salt. The package of interventions will involve patients receiving text messages, telephone calls, emails and written information. They will complete a questionnaire and collect urine samples which will can be used to measure the amount of salt that they are eating. No more than 6 visits will be required. The study is funded by the British Renal Society which is a charity that funds research to help patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with CKD and an eGFR ≥ 20 ml/min/1.73m2
* Participant has clinically acceptable laboratory data available to confirm the diagnosis.
* Able (in the opinion of the Investigators) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

* Female participants who is pregnant, lactating or planning pregnancy during the course of the study.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Inability to understand English or special communication needs because the interventions will use English and is not funded to deal with special communication needs.
* Known salt losing nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A O'Callaghan, MD PhD, Principal Investigator — University of Oxford, UK
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] O'Callaghan CA, Camidge C, Thomas R, Reschen ME, Maycock AJ, Lasserson DS, Fox RA, Thomas NPB, Shine B, James T. Evaluation of a Simple Low-cost Intervention to Empower People with CKD to Reduce Their Dietary Salt Intake: OxCKD1, a Multicenter Randomized Controlled Trial. Kidney360. 2023 Jul 1;4(7):890-898. doi: 10.34067/KID.0000000000000160. Epub 2023 May 31. PMID 37254243
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- See also: University of Oxford Department of Medicine website — http://www.ndm.ox.ac.uk
- See also: British Renal Society — http://www.britishrenal.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note. 201 participants were enrolled into the study following informed consent. Following informed consent, there was a 1-month period of normal routine care after which participants reattended and were randomized to the intervention or to normal routine care (the control group). Only 193 participants attended for randomization.
Period: Overall Study
Arm/Group | Intervention | Normal Care
Started | 96 | 97
Completed | 77 | 81
Not Completed | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Normal Care | Total
Number analyzed (Participants) | 96 | 97 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.8) | 64.2 (10.5) | 63.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 47 | 49 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 2 | 0 | 2
  Any other Asian background | 1 | 0 | 1
  Any other ethnic group | 0 | 1 | 1
  Any other mixed background | 1 | 1 | 2
  Any other White background | 5 | 3 | 8
  British | 84 | 86 | 170
  Caribbean | 0 | 2 | 2
  Irish | 2 | 2 | 4
  Pakistani | 1 | 0 | 1
  White and Asian | 0 | 1 | 1
  White and Black African | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 96 | 97 | 193
24-hour urinary sodium excretion [Mean (Standard Deviation); unit: mmol/day] | 125 (53) | 134 (58) | 129 (56)
24-hour urinary salt excretion [Mean (Standard Deviation); unit: grams/ day] | 7.3 (3.1) | 7.8 (3.4) | 7.6 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Urinary Sodium Excretion
Description: To evaluate whether a new care bundle helps patients to reduce their salt intake.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Intervention | Normal Care
Number analyzed (Participants) | 77 | 81
mmol/day | 93 (48) | 119 (52)

2. Primary Outcome: 24-hour Urinary Salt Excretion
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: grams/ day
Arm/Group | Intervention | Normal Care
Number analyzed (Participants) | 77 | 81
grams/ day | 5.4 (2.8) | 6.9 (3.1)

3. Secondary Outcome: 24-hour Urinary Sodium Excretion
Time Frame: 3 months
Population: The primary study period was 1 month after randomization to the intervention or to normal routine care (the control group). Participants were invited to further assessment 3 months following randomization and 69 in the control group and 65 in the intervention group undertook this.
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Intervention | Normal Care
Number analyzed (Participants) | 65 | 69
mmol/day | 100 (41) | 113 (52)

4. Secondary Outcome: 24-hour Urinary Salt Excretion
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams/ day
Arm/Group | Intervention | Normal Care
Number analyzed (Participants) | 65 | 69
grams/ day | 5.9 (2.4) | 6.6 (3.1)

5. Secondary Outcome: 24-hour Urinary Sodium Excretion
Time Frame: 11 months
Population: The primary study period was 1 month after randomization to the intervention or to normal routine care (the control group). Participants were invited to further assessment 11 months following randomization and 16 in the control group and 44 in the intervention group undertook this.
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Intervention | Normal Care
Number analyzed (Participants) | 44 | 16
mmol/day | 106 (41) | 121 (58)

6. Secondary Outcome: 24-hour Urinary Salt Excretion
Time Frame: 11 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams/ day
Arm/Group | Intervention | Normal Care
Number analyzed (Participants) | 44 | 16
grams/ day | 6.2 (2.4) | 7.1 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the primary study period which was from the date of consent to the end of the one month period during which participants were either randomized to the intervention or to normal routine care (the control group). Further adverse event data was also collected from those participants who attended for further invited assessments at 3 or 11 months following randomization.
Arm/Group | Intervention | Normal Care
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/97
Other Adverse Events (participants affected / at risk) | 0/96 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No